CLINICAL TRIAL: NCT05848362
Title: Comparison of Blood Glucose Measurement Values Taken by Different Methods in Intensive Care Unit (ICU) Patients
Brief Title: Comparison of Blood Glucose Measurement Values
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Hulya Yilmaz, Pirincipal Investigator, PhD, Msc, Uludag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16/03/2022 - 6/10
Record Dates: First submitted 2023-04-05; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Pain, Acute; Glucose Test Site Bleeding
Keywords: blood glucose measurements; intensive care patients; venous blood; capillary blood; arterial blood
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental study with a single group and simultaneous (matched) sample will conduct with the purpose of to determine whether glucose values are different for a bedside glucose meter compared to the main clinical laboratory and whether the blood sampling site has a significant effect on glucose values.
Masking Description: single group sample, there is no blinding as everyone will be treated equally
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SINGLE GROUP (Other): This is a quasi-experimental study with a single group and simultaneous (matched) sample will conduct with the purpose of to determine whether glucose values are different for a bedside glucose meter compared to the main clinical laboratory and whether the blood sampling site has a significant effect on glucose values.
  Interventions: Other: Blood Glucose Measurement Values Taken by Different Methods

INTERVENTIONS:
Other: Blood Glucose Measurement Values Taken by Different Methods — In total, blood samples will be collected from 3 different sites (central venous catheter, capillary, arterial catheterization) in the same patient. In total, with 5 different techniques from 3 different regions from the same patient;
  ARTERIAL BLOOD SAMPLE i) Washing with 5 cc 1% Heparin fluid ii) Washing with 10 cc 1% Heparin fluid CAPILAR BLOOD SAMPLE iii) Right / Left Fingertip iv) Thumb base CENTRAL VENOUS CATHETERIZATION BLOOD SAMPLE will be collected.

SUMMARY:
Purpose: It is one of the important nursing interventions for patients in intensive care units with strict glycemic protocol to determine whether glucose values are different for a bedside glucose meter compared to the main clinical laboratory and whether the blood sampling site has a significant effect on glucose values. In this study, it is aimed to compare whether there is a difference between blood samples from venous, arterial, capillary and thumb base region, which is defined as an alternative region to the fingertip, in blood glucose level measurement, and to compare the consistency between the thumb base region and fingertip region and pain and results of the different methods used.

Methods: The universe of the research consists of Bursa Uludağ University Health Practice and Patients will be hospitalized in the General Surgery Intensive Care Unit of the Research Center between April and September 2023. 125 patients who meet the sample selection criteria will form the sample of the study. The sample size of the study was determined statistically with the G*Power (3.1.7) program. Comparison of blood glucose measurement taken with different methods in the power analysis to determine the sample size. When the effect size of blood glucose was determined as 0.9, it was calculated that a total of 125 patients should be included for a significance level of 0.05 and a power of 80%. Research '' Ergin E., Zaybak A. (2022). Effects of different methods used to take blood samples on blood glucose measurements. Reference is made to Clinical Nursing Research, 31(1), (p.29-38).DOI: 10.1177/10547738211024782". 125 patients who meet the sample selection criteria will form the sample of the study. The sample size of the study was determined statistically with the G*Power (3.1.7) program. When the effect size of blood glucose was determined as 0.9 in the comparison of blood glucose measurement taken with different methods in the power analysis performed to determine the sample size, it was calculated that a total of 125 patients should be included for a significance level of 0.05 and a power of 80%.

DETAILED DESCRIPTION:
Purpose: In this study, it is aimed to compare whether there is a difference between blood samples from venous, arterial, capillary, and thumb base regions, which is defined as an alternative region to the fingertip, in blood glucose level measurement, and to compare the consistency between the thumb base region and fingertip region and pain and results of the different methods used.

Design: This is a quasi-experimental study with a single group and simultaneous (matched) sample will conduct to determine whether glucose values are different for a bedside glucose meter compared to the main clinical laboratory and whether the blood sampling site has a significant effect on glucose values.

A central venous catheter blood sample will be taken from the patient by the guideline recommendations and placed in the biochemistry tube and taken to the laboratory by the researchers. This result is studied by the "biochemistry-glucose test" laboratory.

A capillary blood sample (right/left fingertip; thumb base) from the same patient will be evaluated with a glucometer (Accu-check).

Finally, from the same patient, the transducer set to which the arterial catheterization is connected will first be washed with 5 ccs 1% heparin, and blood glucose will be measured by taking a blood sample from the catheter. Then, it will be washed with 10 ccs 1% heparin and a blood sample will be taken from the catheter and blood glucose measurement will be made. An arterial blood sample (right/left fingertip; thumb base) from the same patient will be evaluated with a glucometer (Accu-check).

The purpose of examining this difference is whether a routine transduce set washing has an effect on blood glucose measurement in blood samples taken from patients with arterial catheterization. In total, blood samples will be collected from 3 different sites (central venous catheter, capillary, and arterial catheterization) in the same patient. In total, with 5 different techniques from 3 different regions of the same patient;

ARTERIAL BLOOD SAMPLE i) Washing with 5 ccs 1% Heparin fluid ii) Washing with 10 ccs 1% Heparin fluid CAPILAR BLOOD SAMPLE iii) Right / Left Fingertip iv) Thumb base CENTRAL VENOUS CATHETERIZATION BLOOD SAMPLE will be collected.

ELIGIBILITY:
Inclusion Criteria:

* patients who age bigger than18
* patients who have capillary fullness is good
* patients who have a central venous catheter
* patients who have an arterial catheter

Exclusion Criteria:

* patients who have predibatic will be excluded from the study. The research has been added to the exclusion criteria and has been changed both in the relevant field in the system and in the project application file. In the ADA (American Diabetes Association) definition of prediabetes, IGT (Impaired Glucose Tolerance) (140-200 mg/dl), lower IAG (Impaired Fasting Glucose) (100-125 mg/dl) and additional supplementation according to WHO (World Health Organization) It is based on the criteria of hemoglobin A1c (HbA1c: Hemoglobin A1c) between 5.7% and 6.4% (ADA,2014). Meeting one of the three criteria is defined as prediabetes. Prediabetes screening is performed using 75 g OGTT, HbA1C, FPG, or a 2-hour oral glucose challenge test.
* patients with Diabetes Mellitus,
* patients with coagulopathy
* patients who receive high-dose vasopressors, acetamifon, ascorbic acid, mannitol, corticosteroid, renal replacement therapy
* patients who do not agree to participate in the research,
* patients who have upper extremity amputation, cast, etc. (capillary blood sample cannot be taken for reasons)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2023-05-17 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose Measurement | baseline
  In this comparison, the central venous catheter blood glucose measurement value will be taken as a baseline.

SECONDARY OUTCOMES:
Behavioral Pain Scale | through study completion, an average of 1 year
  The behavioral pain scale consists of three main variables including facial expression, upper extremity, and compliance with the ventilator. An increase in the obtained score indicates an increase in the level of pain. The first items in each sub-dimension describe the absence of pain, the second items describe mild, the third items moderate, and the fourth items describe increased pain levels. Each sub-dimension is scored between 1 (no response to pain) and 4 (complete response to pain). The lowest score obtained from the scale is 3 and the highest score is 12. As the score increases, the level of pain increases. The first items indicate no pain, the second items indicate mild pain, the third items indicate the presence of moderate pain, and the fourth items indicate the presence of severe pain. The behavioral pain scale has been proven to be valid and reliable for assessing pain in intubated patients in the ICU.
Visual Analog Scale | through study completion, an average of 1 year
  It is a one-dimensional scale used in the measurement of VAS pain. Among the one-dimensional scales used to determine the severity of pain in patients, it was determined that the VAS measures more sensitively and is more reliable. The scale consists of a 100 mm long horizontal line. On one end are the phrases "No Pain" and on the other end "Unbearable Pain" describing the most severe pain possible. The patient is asked to mark his pain on the scale. The length of the line from the starting point of the scale to the point marked by the patient is measured and recorded in mm. After capillary blood glucose measurement is made, the patients will be educated by the researcher about the use of VAS before the research and the patients will be asked to evaluate their pain using VAS. It will be recorded in the data collection form as the numerical value obtained by measuring the point where the patient marked on the scale.

IPD SHARING:
Plan to Share IPD: No
No Individual participant data (IPD) doesn't share any other researchers. Only research team will see data on IPD. After the data collection phase is completed and turned into a publication, other researchers can access the publication.

REFERENCES:
- [Background] Payen JF, Bru O, Bosson JL, Lagrasta A, Novel E, Deschaux I, Lavagne P, Jacquot C. Assessing pain in critically ill sedated patients by using a behavioral pain scale. Crit Care Med. 2001 Dec;29(12):2258-63. doi: 10.1097/00003246-200112000-00004. PMID 11801819
- [Background] Pinheiro ARPQ, Marques RMD. Behavioral Pain Scale and Critical Care Pain Observation Tool for pain evaluation in orotracheally tubed critical patients. A systematic review of the literature. Rev Bras Ter Intensiva. 2019 Oct-Dec;31(4):571-581. doi: 10.5935/0103-507X.20190070. PMID 31967234
- [Background] Hirose T, Mita T, Fujitani Y, Kawamori R, Watada H. Glucose monitoring after fruit peeling: pseudohyperglycemia when neglecting hand washing before fingertip blood sampling: wash your hands with tap water before you check blood glucose level. Diabetes Care. 2011 Mar;34(3):596-7. doi: 10.2337/dc10-1705. Epub 2011 Jan 31. PMID 21282342
- [Background] Rabinstein AA. Hyperglycemia in critical illness: lessons from NICE-SUGAR. Neurocrit Care. 2009;11(1):131-2. doi: 10.1007/s12028-009-9240-x. Epub 2009 Jun 5. No abstract available. PMID 19499351
- [Background] Ergin E, Zaybak A. Effects of Different Methods Used to Take Blood Samples on Blood Glucose Measurements. Clin Nurs Res. 2022 Jan;31(1):29-38. doi: 10.1177/10547738211024782. Epub 2021 Jul 5. PMID 34218680